CLINICAL TRIAL: NCT00908323
Title: Characterization of the Innate Immune Response to Candidate HIV Vaccines, an Ancillary Study to HVTN 205
Brief Title: Early Immune Responses to Vaccination - A Substudy to HVTN 205
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HVTN 908; 10806 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples 30 - 90 mL per visit

GROUPS / COHORTS (2):
- A: Participants receiving the JS7 DNA and MVA/HIV62 vaccinations in HVTN 205
  Interventions: Biological: JS7 DNA vaccine; Biological: MVA/HIV62 vaccine
- B: Participants receiving the placebos of the JS7 DNA and MVA/HIV62 vaccines in HVTN 205
  Interventions: Biological: JS7 DNA vaccine; Biological: MVA/HIV62 vaccine

INTERVENTIONS:
Biological: JS7 DNA vaccine
Biological: MVA/HIV62 vaccine

SUMMARY:
HVTN 908 is a sub study of the HIV vaccine trial, HVTN 205. The purpose of this sub study is to better understand how a person's immune system responds to vaccines, particularly HIV vaccines. More specifically, researchers will determine whether early responses in the immune system help predict strong and long-lasting immunity.

DETAILED DESCRIPTION:
Some of the first HIV vaccines were designed to trigger neutralizing antibody responses as a way to prevent HIV infection. Unfortunately, the first versions of these vaccines were not able to achieve their desired response. An alternative strategy to the antibody approach is the stimulation of HIV-specific CD8 T-lymphocyte (CTL) responses. CTL responses were previously demonstrated to play an important role in the control of simian immunodeficiency virus (SIV), the HIV equivalent studied in rhesus macaque monkeys. Additionally, other studies suggest CTLs play an important role in viral control during chronic infection. Based on this information, several groups have shifted their focus to the development of CTL-based vaccines, some of which have entered advanced clinical trials.

A DNA/rMVA vaccine strategy is structured to bring about both T cell and antibody responses. The primary vaccination is DNA based and will express only HIV proteins as a way to produce an HIV-focused immune response. A secondary, rMVA boost vaccination, which expresses both HIV and MVA proteins will ideally amplify the focused response of the initial vaccination. The DNA and rMVA are physically two different vaccinations given at separate times but together they make up one preventive regimen. Both vaccine components express non-infectious virus-like particles.

The main study, HVTN 205 will evaluate the safety of and immune response to a two vaccine regimen in healthy, HIV-uninfected adults who never received an HIV preventive vaccine before. HVTN 205 will include two parts, Part A, in which the two vaccine regimen is compared to a placebo, and Part B, in which the two vaccine regimen will be compared to both a placebo and a single vaccine regimen with the rMVA vaccine.

HVTN 908 is a sub study of HVTN 205, and will explore the innate immune response to candidate HIV vaccines. In particular, researchers will study whether early immune response following vaccination can predict strong and long-lasting immunity. They will also study whether varying types of vaccines promote different immune responses soon after vaccination.

Only participants enrolled in HVTN 205 are eligible for HVTN 908. Approximately 50 participants will be recruited for the duration of 12 months per participant. The study will last for a total of 2 years, including enrollment, follow-up, and analysis. Potential participants of the sub study will undergo a screening visit before eligibility can be determined. Screening may involve a physical exam, health history, and blood tests.

There will be some additional visits for participants of HVTN 908 that are not included in the main study. Some main study visits may also take extra time for participants enrolled in the sub study. Blood samples will be taken at study visits. These samples are taken in addition to those for the main study.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled receipt of a vaccine or placebo in HVTN 205
* For participants in Part B of HVTN 205, enrollment in HVTN 908 and HVTN 205 at the same time
* HVTN 908 assessment of understanding: completion of a questionnaire prior to enrollment; demonstration of understanding for all questionnaire items answered incorrectly.
* Body weight of 50 kg (110 lbs) or more
* Hemoglobin of 12.0 g/dL or more for female volunteers, and 13.0 g/dL or more for male volunteers
* Negative HIV-1 and -2 blood test

Exclusion Criteria:

* Clinically significant medical condition, physical examination finding, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the study protocol.
* Any medical, psychiatric, or occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, or a participant's ability to give informed consent
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants enrolled in HVTN 205
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of lymphocyte populations, dendritic cells, monocytes, and granulocytes | Throughout study
Serum concentrations of cytokines and chemokines | Throughout study
Changes in PBMC gene expression relative to prevaccine levels of key genes expected to change, such as IP-10 and MCP-1 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Erica Andersen-Nissen, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Baker BM, Block BL, Rothchild AC, Walker BD. Elite control of HIV infection: implications for vaccine design. Expert Opin Biol Ther. 2009 Jan;9(1):55-69. doi: 10.1517/14712590802571928. PMID 19063693
- [Background] Browne EP, Littman DR. Myd88 is required for an antibody response to retroviral infection. PLoS Pathog. 2009 Feb;5(2):e1000298. doi: 10.1371/journal.ppat.1000298. Epub 2009 Feb 13. PMID 19214214
- [Background] Zwolinska K. [Host genetic factors associated with susceptibility to HIV infection and progression of infection]. Postepy Hig Med Dosw (Online). 2009 Feb 24;63:73-91. Polish. PMID 19252466